CLINICAL TRIAL: NCT05113238
Title: Oocyte Activation: Revised or Initial Activated Gamete Treatment (AGT) Technique, Which is Better?! A Sibling-oocytes-split Design and Case Series of Chemical Pregnancies
Brief Title: Oocyte Activation: Revised or Initial AGT Technique, Which is Better?! A Sibling-oocytes-split Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Fertility Center, Egypt (Other)
Collaborators: Hawaa Fertility Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 003
Record Dates: First submitted 2021-10-08; First posted 2021-11-09 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Assisted Reproductive Technology
Keywords: Calcium ionophore; gamete activation; ICSI; male factor

STUDY DESIGN:
Intervention Model Description: single group of patients will be conducted into sibling-oocyte-split design
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AGT-Initial (Active Comparator): Oocytes will be injected with spermatozoa and will be incubated in 10 mM calcium ionophore (Sigma-Aldrich) for two rounds of 10 minutes at 37 C, 30 minutes after ICSI injection, and then will be rinsed and transferred into culture medium.
  Interventions: Procedure: Assisted gamete activation
- AGT-revised (Experimental): ejaculated spermatozoa will be exposed to calcium ionophore in a drop on the ICSI dish before injection. During the ICSI procedure, spermatozoa will be aspirated individually from the drop containing calcium ionophore and immobilized in a separate PVP drop. Next, approximately 0.4 pL of calcium ionophore will be aspirated into the micropipette and injected into the oocyte with the spermatozoa.
  Post-ICSI oocytes will be then exposed to 50 mM calcium ionophore for 10 minutes at 37C, and then will be washed and placed in culture medium.
  Interventions: Procedure: Assisted gamete activation

INTERVENTIONS:
Procedure: Assisted gamete activation — compare two different assisted gamete activation protocols to improve ICSI outcome

SUMMARY:
This study will be conducted to compare two different Assisted Gamete treatment (AGT) with oocyte-sibling-split design control group : AGT- initial protocol for activating oocytes by culturing oocytes in calcium ionophore after injection for two rounds of 10 minutes at 37 C, 30 minutes after injection.

sample group : AGT-revised protocol oocytes will be injected by sperm previously cultured in Ca ionophore and 0.4 pL of calcium ionophore then will be cultured in calcium ionophore after injection for 10 minutes

DETAILED DESCRIPTION:
investigators performed ICSI then with one of two activation protocols added : AGT-initial or AGT-revised For the AGT initial protocol, Oocytes will be injected then will be incubated in 10 mM calcium ionophore (Sigma-Aldrich) for two rounds of 10 minutes at 37 C, 30 minutes after ICSI injection, and then will be rinsed and transferred into culture medium.

For the AGT-revised protocol, ejaculated spermatozoa will be exposed to calcium ionophore in a drop on the ICSI dish before injection. During the ICSI procedure, spermatozoa will be aspirated individually from the drop containing calcium ionophore and immobilized in a separate polyvinylpyrrolidone drop. Next, approximately 0.4 pL of calcium ionophore will be aspirated into the micropipette and will be injected into the oocyte with the spermatozoa. Post-ICSI oocytes will be then exposed to 50 mM calcium ionophore for 10 minutes at 37 C, and then will be washed and placed in culture medium.

ELIGIBILITY:
Inclusion Criteria:

* couples presented with an extremely poor fertilization (<10%)
* couples with previous complete fertilization failure after undergoing ICSI cycles
* At least 4 MII oocytes
* Severe oligoasthinozoospermia
* Teratozoospermia
* testicular aspirated sperm

Exclusion Criteria:

* age >40 years
* BMI >34
* aspirated oocytes < 4
* Normozoospermia
* subfertile patients

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 222 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2021-12-25 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Number of top quality day 3 embryos | 3 days after ICSI procedure day
  number of top quality embryos
Number of Top quality day 4 embryos | 4 days after ICSI procedure
  number of top quality embryos
Number of Top quality day 5 embryos | 5 days after ICSI procedure
  number of top quality embryos

SECONDARY OUTCOMES:
chemical pregnancy rate | 15 days after embryo transfer procedure day
  the number of positive pregnancy cases from overall cases

CONTACTS AND LOCATIONS:
Overall Officials: Sahar SA Eissa, PHD, Study Director — research team leader; Engy EA Abdallah, M.sc, Study Chair — investigator & researcher
Locations (1):
- Royal Fertility Center, Al Mansurah, Daqahlya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study protocol and outcome
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: two months